CLINICAL TRIAL: NCT03070665
Title: Increasing Blood Pressure During Gastric ESD May Control the Risk of Postoperative Bleeding: a Prospective Randomized Trial
Brief Title: Blood Pressure During ESD is Related With the Postoperative Bleeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: ZS-GI
Record Dates: First submitted 2017-02-23; First posted 2017-03-03 (Actual); Last update posted 2017-04-26 (Actual); Status verified 2017-03

CONDITIONS: Gastrointestinal Disease; Gastrointestinal Bleeding
Keywords: endoscopic submucosal dissection; postoperation bleeding
MeSH Terms: conditions — Gastrointestinal Diseases; Gastrointestinal Hemorrhage | interventions — Norepinephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Increasing blood pressure (Experimental): Using norepinephrine pump as the initial dose is 0.05μg/Kg.min to increase the patient's blood pressure up to about 150 mmHg for 5 min during ESD.
  Interventions: Drug: Norepinephrine
- Control group (No Intervention): Patients received normal ESD manipulation.

INTERVENTIONS:
Drug: Norepinephrine — Increasing blood pressure up to 150mmHg for 5min using norepinephrine pump as initial dose 0.05μg/Kg.min during ESD operation, meanwhile check out the potential hemorrhage spot which is not obvious and then use the hot biopsy forceps to coagulate the bleeding spot, after that withdraw the norepinephrine and record the potential bleeding spot's location. The other procedures are the same as control groups'.
  Other Names: ephedrine; phenylephedrine
  Arms: Increasing blood pressure

SUMMARY:
Endoscopic submucosal dissection(ESD) is a prominent minimally invasive operation technique for treating early gastrointestinal tumor. But promoting ESD is uneasy because of its complications such as postoperative bleeding, perforation and so on. So if we decrease the rate of postoperative bleeding, ESD might be better popularized. Some study indicated that hypertension was the independent risk factor of postoperative bleeding. Endoscopic center of Fudan University Zhongshan Hospital is a rich experienced medical unit in doing ESD operation in China. Referring to our experience, if we can use some special methods to find the potential bleeding spot which is not obvious during ESD operation and we coagulate it precisely, then we may control the risk of postoperative bleeding.

Based on the above hypothesis, our team designed this study to examine whether increasing blood pressure during gastric ESD could help to control the risk of postoperative bleeding.

ELIGIBILITY:
Inclusion Criteria:

* A. The indications for ESD for gastric neoplasms, such as intramucosal gastric cancer and adenoma, include intramucosal differentiated tubular adenocarcinoma of any size without ulceration or signs of submucosal invasion and intramucosal differentiated-type adenocarcinoma of less than 3 cm with an ulcer scar. The histology, tumor location, and depth of invasion fulfilled the criteria of the Japanese Research Society for Gastric Cancer.

B. The eligible patients' blood coagulation function should be normal without any associated medicine influenced.

Exclusion Criteria:

* A. Previously treated by radical gastrectomy. B. Pregnant or on breast feeding. C. Patients who are unwilling or unable to provide informed consent, such as those with psychiatric problem, drug abuse or alcoholism.

D. Coagulopathy: liver cirrhosis, thrombocytopenia. E. Anti-platelet agents. Allergic to PPI or norepinephrine. F. Patients with sever hypertension(systolic pressure>180mmHg), or the hypotensor cann't control blood pressure suitably.

G. Patients with cardiovascular and cerebrovascular events within 6 months.

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 296 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
PostESD bleeding | 60 days
  Post-ESD bleeding was defined as clinical evidence of bleeding after ESD, manifesting as hematemesis or melena, which required urgent endoscopic treatment

SECONDARY OUTCOMES:
Post-ESD perforation | 60 days
  Post-ESD perforation was defined as the clinical symptoms such as abdominal pain, abdominal distension, fever and so on, then combined abdominal CT images.
Hospitalization | 60 days
  length of stay in hospital
Post-ESD hemoglobin | 60 days
  The patient's postoperative hemoglobin will be examined 24-48h after ESD operation, and will be analyzed by the software of SPSS19.0 compared with the figure of pre-operation.
Post-ESD hemocrit | 60 days
  The patient's postoperative hemocrit will be examined 24-48h after ESD operation, and will be analyzed by the software of SPSS19.0 compared with the figure of pre-operation.
Post-ESD prothrombin time | 60 days
  The patient's postoperative prothrombin time will be tested 24-48h after ESD operation, and will be analyzed by the software of SPSS19.0 compared with the figure of pre-operation.
Post-ESD activated partial prothrombin time | 60 days
  The patient's postoperative activated partial prothrombin time will be tested 24-48h after ESD operation, and will be analyzed by the software of SPSS19.0 compared with the figure of pre-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Zhou Pinghong, Doctor, Study Director — Shanghai Zhongshan Hospital of Fudan University
Locations (1):
- Zhongshan Hospital, Shanghai, SHA, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ebi M, Shimura T, Nishiwaki H, Tanaka M, Tsukamoto H, Ozeki K, Sawada T, Mizoshita T, Mori Y, Kubota E, Tanida S, Kataoka H, Joh T. Management of systolic blood pressure after endoscopic submucosal dissection is crucial for prevention of post-ESD gastric bleeding. Eur J Gastroenterol Hepatol. 2014 May;26(5):504-9. doi: 10.1097/MEG.0000000000000072. PMID 24589830
- [Background] Watari J, Tomita T, Toyoshima F, Sakurai J, Kondo T, Asano H, Yamasaki T, Okugawa T, Ikehara H, Oshima T, Fukui H, Miwa H. Clinical outcomes and risk factors for perforation in gastric endoscopic submucosal dissection: A prospective pilot study. World J Gastrointest Endosc. 2013 Jun 16;5(6):281-7. doi: 10.4253/wjge.v5.i6.281. PMID 23772265
- [Background] Kim JS, Chung MW, Chung CY, Park HC, Ryang DY, Myung DS, Cho SB, Lee WS, Joo YE. The need for second-look endoscopy to prevent delayed bleeding after endoscopic submucosal dissection for gastric neoplasms: a prospective randomized trial. Gut Liver. 2014 Sep;8(5):480-6. doi: 10.5009/gnl13226. Epub 2014 Feb 24. PMID 25228971
- [Background] Morgenstern LB, Demchuk AM, Kim DH, Frankowski RF, Grotta JC. Rebleeding leads to poor outcome in ultra-early craniotomy for intracerebral hemorrhage. Neurology. 2001 May 22;56(10):1294-9. doi: 10.1212/wnl.56.10.1294. PMID 11376176
- [Background] Ryu SJ, Kim BW, Kim BG, Kim JH, Kim JS, Kim JI, Park JM, Oh JH, Kim TH, Kim JJ, Park SM, Park CH, Song KY, Lee JH, Kim SG, Kim DJ, Kim W. Endoscopic submucosal dissection versus surgical resection for early gastric cancer: a retrospective multicenter study on immediate and long-term outcome over 5 years. Surg Endosc. 2016 Dec;30(12):5283-5289. doi: 10.1007/s00464-016-4877-y. Epub 2016 Jun 23. PMID 27338583
- [Background] Jang JS, Choi SR, Graham DY, Kwon HC, Kim MC, Jeong JS, Won JJ, Han SY, Noh MH, Lee JH, Lee SW, Baek YH, Kim MJ, Jeong DS, Kim SK. Risk factors for immediate and delayed bleeding associated with endoscopic submucosal dissection of gastric neoplastic lesions. Scand J Gastroenterol. 2009;44(11):1370-6. doi: 10.3109/00365520903194609. PMID 19891589
- [Background] Suzuki S, Chino A, Kishihara T, Uragami N, Tamegai Y, Suganuma T, Fujisaki J, Matsuura M, Itoi T, Gotoda T, Igarashi M, Moriyasu F. Risk factors for bleeding after endoscopic submucosal dissection of colorectal neoplasms. World J Gastroenterol. 2014 Feb 21;20(7):1839-45. doi: 10.3748/wjg.v20.i7.1839. PMID 24587661